CLINICAL TRIAL: NCT05759429
Title: Effect of Melatonin on Oxidative Stress in Obese Adults Undergoing an Acute Exercise Session
Brief Title: Effect of Melatonin on Oxidative Stress in Obese Adults (MELASTRESSOB)
Acronym: MELASTRESSOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01C127
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Obesity; Melatonin; Oxidative stress; Adulthood
MeSH Terms: conditions — Obesity | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated multidisciplinary body weight reduction program (BWRP) (Active Comparator)
  Interventions: Other: BWRP
- Integrated multidisciplinary body weight reduction program (BWRP) + melatonin (Active Comparator)
  Interventions: Other: BWRP + melatonin

INTERVENTIONS:
Other: BWRP — Physical exercise protocol after 1 and 15 days of integrated multidisciplinary BWRP, which includes a low-calorie diet, physical activity, psychological support, and nutritional education
  Arms: Integrated multidisciplinary body weight reduction program (BWRP)
Other: BWRP + melatonin — Physical exercise protocol after 1 and 15 days of integrated multidisciplinary BWRP and melatonin (4 mg/die), administered 2-3 hours before bedtime
  Arms: Integrated multidisciplinary body weight reduction program (BWRP) + melatonin

SUMMARY:
The present research project aims to evaluate oxidative stress in a cohort of obese adults, subjected to an in-hospital 3-week multidisciplinary body weight reduction program (BWRP) with or without melatonin. Our hypothesis is that melatonin, administered to the obese subject, could be effective in reducing the oxidative stress associated with physical exercise (acute).

Specifically, the main objective will be to investigate a difference in the mean levels of some peripheral oxidative stress markers at their peak during an acute exercise session in the two groups (primary endpoint).

Secondly, the possible pre-post difference (baseline vs end of treatment) of the peak of each oxidative stress marker between the two groups will be evaluated (secondary endpoint

DETAILED DESCRIPTION:
Materials and methods 20 obese subjects (F/M = 10/10; age range 18-40 years; body mass index, BMI > 30 kg/m2), hospitalized for a period of integrated metabolic rehabilitation (BWRP) at the Division of Metabolic Diseases, Istituto Auxologico Italiano, Piancavallo (VB), Italy.

After verifying the inclusion/exclusion criteria, including the absence of other relevant pathologies apart from obesity, we will proceed with the collection of clinical data (heart rate, blood pressure, body temperature) and anthropometric data (weight, height, BMI, waist circumference, hip circumference), including assessment of body composition with bio-impedancemetry.

According to a randomized scheme, with the only constraint of maintaining a 1/1 ratio for sex, the subjects will undergo one of the following interventions:

1. Integrated multidisciplinary BWRP, which includes a low-calorie diet, physical activity, psychological support, and nutritional education;
2. Integrated multidisciplinary BWRP (as above) combined with melatonin. Melatonin will be administered during 15 consecutive days of our standard BWRP, after dinner, and 2-3 hours before bedtime. The first dose will be administered on the same evening of the day in which the incremental exercise (test 1, baseline G0) will be performed, necessary to establish the execution conditions of test 2.

The acute exercise session (test 2, described below) will be performed at D1 and D15 (days 1-15 of BWRP).

Each subject will conduct the following exercise protocols:

1. Incremental exercise (4 min rest, 3 min walk at 4 km/h and 0% incline followed by 1% incline and speed increments of 0.5 km/h every minute), breathing a mixture composed of 21 % O2 in nitrogen (ambient air, O2-N2); this exercise is necessary to establish the execution conditions of test 2, which represents the effective exercise that will be performed before and after the intervention and during which the blood samples described below will be taken;
2. Moderate intensity constant load exercise, at a load corresponding to 60% of the aerobic threshold, determined during the above incremental exercise, conducted for 30 minutes or until voluntary exhaustion, performed at D1 and D15.

All tests will be monitored and supervised by dedicated personnel. For each of the two acute exercise sessions (i.e., before starting the BWRP-G1 and after the BWRP-G15 intervention), four blood draws will be taken: in baseline conditions (pre-exercise), immediately at the end of the 'exercise, and 60-120 minutes after the end of exercise (T0', T30', T90' and T150', respectively), to identify the peak of each marker.

In plasma/serum samples taken basally (T0'), at the end of exercise (T30'), 60' post (T90'), and 120' post (T150') after the end of the exercise, a panel of markers will be determined peripheral oxidative stress. In particular:

* dROMS (reactive oxygen species)
* MDA (malondialdehyde)
* Oxidized/reduced GSH (glutathione).
* FRAP (plasma iron-reducing capacity, which corresponds to the total antioxidant capacity);
* melatonin and tryptophan metabolites. TNF-α, IL-6, and IL-8 levels will be determined in plasma/serum samples taken basally (T0') and at the end of physical exercise (T30'). Finally, the basal glucometabolic profile (glucose, insulin, HOMA-IR, glycated Hb, triglycerides, total cholesterol, LDL, HDL, and hsPCR) will be analyzed in the basal plasma/serum samples (T0').

Approval of the protocol by the Ethics Committee will be required; informed consent will be collected from all participants.

ELIGIBILITY:
Inclusion Criteria:

* body mass index > 30 kg/m2
* absence of concomitant relevant diseases, apart severe obesity
* hospitalized for a period of integrated metabolic rehabilitation

Exclusion Criteria:

- concomitant relevant diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
dROMS (reactive oxygen species) during physical exercise protocol | Baseline (T0'), after 30 minutes of the physical exercise protocol (T30') and at T90' and T120' at day 1 and day 15 of the intervention
  Change in dROMS
Malondialdehyde (MDA) during physical exercise protocol | Baseline and after 30, 60, 90 and 120 minutes of the physical exercise protocol at day 15 of the intervention
  Change in malondialdehyde
Ratio of oxidized/reduced GSH (glutathione) during physical exercise protocol | Baseline (T0'), after 30 minutes of the physical exercise protocol (T30') and at T90' and T120' at day 1 and day 15 of the intervention
  Change in ratio of oxidized/reduced GSH (glutathione)
Plasma iron-reducing capacity (FRAP) during physical exercise protocol | Baseline (T0'), after 30 minutes of the physical exercise protocol (T30') and at T90' and T120' at day 1 and day 15 of the intervention
  Change in plasma iron-reducing capacity (FRAP)

SECONDARY OUTCOMES:
Melatonin concentration | Baseline (T0') and after 30 minutes of the physical exercise protocol (T30') at day 1 and day 15 of the intervention
  Change in melatonin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sartorio, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy